CLINICAL TRIAL: NCT04751526
Title: A Non-invasive Intervention (BreEStim) for Management of Phantom Limb Pain (PLP) After Limb Amputation
Brief Title: A Non-invasive Intervention (BreEStim) for Management of Phantom Limb Pain (PLP) After Limb Amputation (Experiment 3)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sheng Li, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-20-1032 (Experiment 3)
Record Dates: First submitted 2021-02-10; First posted 2021-02-12 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Pain Management
Keywords: Phantom Limb Pain; BreEStim
MeSH Terms: conditions — Agnosia; Phantom Limb

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- BreEStim 240, then EStim 240 (Experimental): BreEStim is voluntary breathing controlled transcutaneous electrical nerve stimulation.
  Interventions: Device: BreEStim 240; Device: EStim 240
- EStim 240, then BreEstim 240 (Experimental): EStim is transcutaneous electrical nerve stimulation.
  Interventions: Device: BreEStim 240; Device: EStim 240

INTERVENTIONS:
Device: BreEStim 240 — 240 BreEStim stimuli/visit will be applied for 10 sessions to test any accumulated analgesic effect.
Device: EStim 240 — 240 EStim stimuli/visit will be applied for 10 sessions to test any accumulated analgesic effect.

SUMMARY:
The purpose of this study is to compare the effectiveness of innovative intervention of breathing controlled electrical stimulation (BreEStim) and conventional electrical stimulation (EStim) in management of neuropathic phantom limb pain in patients after limb amputation after multiple sessions of treatment.

DETAILED DESCRIPTION:
Subjects will receive 10-session BreEStim and 10-session EStim treatment in a random order. The interval between BreEStim and EStim is at least 2 weeks. The following assessment will be made before and after

1. Visual analogue scale (VAS).
2. Quantitative sensory testing (QST). It includes non-invasive assessment of tactile sensation threshold (TST), electrical sensation threshold (EST), electrical pain threshold (EPT), and thermal thresholds.
3. Hear rate variability (HRV). It consists of 5-minute electrocardiogram (ECG) recording before and after a treatment session.

ELIGIBILITY:
Inclusion Criteria:

* has phantom limb pain (PLP) after amputation of one limb, upper or lower limb;
* has chronic pain, >3 months;
* is stable on oral pain medications at least two weeks. (patients are allowed to continue their pain medications, i.e., no change in pain medications.)

Exclusion Criteria:

* currently adjusting oral pain medications for their PLP;
* has pain, but not PLP (e.g., from inflammation at the incision wound of the residual limb);
* has a pacemaker, or other metal and/or implanted devices;
* has cognitive impairment from brain injury or are not able to follow commands, or to give consent;
* has amputation in multiple limbs;
* have asthma or other pulmonary diseases;
* are not medically stable;
* have preexisting psychiatric disorders;
* alcohol or drug abuse;
* have a history of seizures/Epilepsy, or taking benzodiazepines, anticonvulsants, and antidepressants.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Li, MD, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (2 Weeks)
Arm/Group | BreEStim 240, Then EStim 240 | EStim 240, Then BreEstim 240
Started | 9 | 9
Completed | 9 | 8
Not Completed | 0 | 1
Period: Washout (About 3 to 12 Months)
Arm/Group | BreEStim 240, Then EStim 240 | EStim 240, Then BreEstim 240
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0
Period: Second Intervention (2 Weeks)
Arm/Group | BreEStim 240, Then EStim 240 | EStim 240, Then BreEstim 240
Started | 4 | 7
Completed | 4 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BreEStim 240, Then EStim 240 | EStim 240, Then BreEstim 240 | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 5 | 14
  >=65 years | 0 | 4 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 8 | 6 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 1 | 4 | 5
  Black or African American | 4 | 3 | 7
  Hispanic or Latino | 3 | 2 | 5
  Asian | 0 | 0 | 0
  Others | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Average Change in Pain as Measured by the Visual Analog Scale (VAS)
Description: VAS Scores are recorded from 0 to 10 with 0 being "no pain" and 10 being "worst pain", a higher score indicating a higher level of pain. For each session change is reported as [(VAS score at baseline) - (VAS Score 10 minutes after each intervention)] - a positive value indicates that the score (and pain level) decreased. For this outcome measure we report the average change over all 10 sessions which is calculated by the sum of all divided by 10.
Time Frame: From Baseline to completion of 10 intervention sessions (about 2 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- BreEStim 240: BreEStim is voluntary breathing controlled transcutaneous electrical nerve stimulation.
  BreEStim 240: 240 BreEStim stimuli/visit will be applied for 10 sessions to test any accumulated analgesic effect.
- EStim 240: EStim is transcutaneous electrical nerve stimulation.
  EStim 240: 240 EStim stimuli/visit will be applied for 10 sessions to test any accumulated analgesic effect.
Arm/Group | BreEStim 240 | EStim 240
Number analyzed (Participants) | 16 | 12
score on a scale | 1.38 (0.69) | 0.93 (0.43)

2. Secondary Outcome: Average Change in Sensation Threshold on Amputated Limb Measured by Electrical Sensation Detection Threshold (EST)
Description: Electrical Sensation Threshold (EST) is the minimum electrical current intensity that a person can reliably perceive as a sensation on their skin. This threshold is self-reported by the subjects, and electrical intensity values are recorded when participants first detect the electrical stimulation.
  For each session change is reported is reported as [(EST at 5 minutes after intervention) - (EST at baseline)] - a positive value indicates a decrease in sensation perception. For this outcome measure we report the average change over all 10 sessions which is calculated by the sum of all divided by 10.
Time Frame: From Baseline to completion of 10 intervention sessions (about 2 weeks)
Measure: Mean (Standard Deviation); unit: mA
Arm/Group | BreEStim 240 | EStim 240
Number analyzed (Participants) | 16 | 12
mA | -0.22 (0.27) | -0.11 (0.37)

3. Secondary Outcome: Average Change in Pain Threshold on Amputated Limb Measured by Electrical Pain Detection Threshold (EPT)
Description: An Electrical Pain Threshold (EPT) refers to the minimum intensity of electrical stimulation required to produce a perceptible pain sensation on a person's skin, essentially measuring the point at which an electrical current becomes painful. The EPT is self-reported by subjects when they feel the electrical intensity begins to cause pain. For each session change is reported as [(EPT at 5 minutes after intervention) - (EPT at baseline)] - a positive value indicates an increase in pain threshold. For this outcome measure we report the average change over all 10 sessions which is calculated by the sum of all divided by 10.
Time Frame: From Baseline to completion of 10 intervention sessions (about 2 weeks)
Measure: Mean (Standard Deviation); unit: mA
Arm/Group | BreEStim 240 | EStim 240
Number analyzed (Participants) | 16 | 12
mA | 3.69 (3.87) | 0.99 (1.51)

4. Other Pre Specified Outcome: Change in Heart Rate Variability (HRV) Measured by Electrocardiogram (ECG)
Description: HRV is a measure of the variation in time between each heartbeat. We use HRV to identify the autonomic nervous system changes after intervention treatment.
Time Frame: Baseline, after 10 intervention sessions, about 2 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 18 months
Arm/Group | BreEStim 240 | EStim 240
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 11/11 | 11/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BreEStim 240 (N=11) | EStim 240 (N=11)
Redness (Skin and subcutaneous tissue disorders) | 1 | 1
Discomfort (Skin and subcutaneous tissue disorders) | 11 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/26/NCT04751526/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT04751526/ICF_001.pdf